CLINICAL TRIAL: NCT07234942
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Single Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7812653 Following Intrathecal Administration in Participants With Early Symptomatic Alzheimer's Disease
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7812653 in Participants With Early Symptomatic Alzheimer's Disease (eAD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP45770; 2025-522101-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RO7812653 (Experimental): Participants will receive a dose of RO7812653
  Interventions: Drug: RO7812653
- Placebo (Placebo Comparator): Participants will receive a dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RO7812653 — Participants will receive RO7812653 as per the schedule in the protocol
  Arms: RO7812653
Drug: Placebo — Participants will receive placebo as per the schedule in the protocol
  Arms: Placebo

SUMMARY:
This study aims to evaluate the safety, tolerability, immunogenicity, pharmacokinetics, and pharmacodynamics following administration of RO7812653 in participants with eAD.

ELIGIBILITY:
Inclusion Criteria:

* Probable AD dementia (consistent with National Institute on Aging and Alzheimer's Association (NIA-AA) core clinical criteria for probable AD dementia) [McKhann et al 2011] or Mild Cognitive Impairment (MCI) due to AD (consistent with the NIA-AA core clinical criteria for mild cognitive impairment due to AD) [Albert et al 2011]).
* Willingness and ability to complete all aspects of the study. The participant should be capable of completing assessments either alone or with the help of the study partner.
* Fluency in the language of the tests used at the study site.
* Adequate visual and auditory acuity, in the investigator's judgment, sufficient to perform the neuropsychological testing (eyewear and hearing aids are permitted).
* If the participant is receiving symptomatic AD medications, a stable dosing regimen for at least 8 weeks prior to screening and until randomization is required.
* Agreement not to participate in other research studies for the duration of this study.

Exclusion Criteria:

* Any medical history or evidence of a condition other than AD that may affect cognition.
* Presence of any significant cerebral abnormalities that would contraindicate lumbar puncture, as assessed on MRI
* Any other significant cerebral abnormalities that the Investigator considers clinically significant
* History of schizophrenia, schizoaffective disorder, major depression or bipolar disorder.'
* Presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological medical conditions which are not stable and adequately controlled or which in the opinion of the investigator could affect the subject's safety in the study or interfere with the study assessments

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2028-04-19 (Estimated); Study Completion 2030-03-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | Up to approximately 40 weeks
Change From Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) Scores | Up to approximately 40 weeks
  C-SSRS measures 4 constructs as follows: severity of ideation, intensity of ideation, behavior, and lethality of actual suicide attempts. Binary (yes/no) data are collected for 10 categories. Numeric ratings are provided for intensity of ideation (if present), from 1 to 5, with 1 being the least severe and 5 being the most severe.

SECONDARY OUTCOMES:
Plasma Concentration of RO7812653 | Up to approximately 40 weeks
Cerebral Spinal Fluid (CSF) Concentration of RO7812653 | Up to approximately 40 weeks
Percentage of Participants with Anti-Drug Antibodies (ADAs) to RO7812653 | Up to approximately 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- National Hospital For Neurology and Neurosurgery, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No